CLINICAL TRIAL: NCT00081848
Title: A Pilot Trial of a CEA-TRICOM Based Vaccine and Radiation to Liver Metastasis in Adults With CEA Positive Solid Tumors
Brief Title: Vaccine Therapy and Radiation to Liver Metastasis in Patients With CEA-Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040167; 04-C-0167; NCT00085241 (obsolete NCT alias)
Record Dates: First submitted 2004-04-22; First posted 2004-04-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-01-25

CONDITIONS: Liver Neoplasms
Keywords: Colon Cancer; Gastrointestinal Cancer; Cytokines; Immunotherapy; Cancer; Solid Tumor; Liver Metastasis
MeSH Terms: conditions — Liver Neoplasms; Colonic Neoplasms; Gastrointestinal Neoplasms; Neoplasms | interventions — Celecoxib

INTERVENTIONS:
Drug: rV-CEA(6D)/TRICOM-rF-CEA(6D)/TRICOM
Drug: rF-CEA(6D)/TRICOM
Drug: Recombinant Fowlpox-GM-CSF
Drug: Celecoxib

SUMMARY:
This study will evaluate the safety and effects of vaccine treatment plus radiation to the liver in patients with solid tumors that have spread to the liver. The vaccine treatment consists of three parts: 1) a "priming vaccine" called rV-CEA(6D)-TRICOM, made from vaccinia virus; 2) a "boosting vaccine" called rF-CEA(6D)-TRICOM), made from fowlpox virus; and 3) a fowlpox virus injected with DNA for GM-CSF, a chemical that boosts the immune system, called rF-GM-CSF. Human DNA is inserted into the priming and boosting vaccine viruses to cause production of proteins that enhance immune activity and also to produce carcinoembryonic antigen (CEA) - a protein that is normally produced by the patient's tumor cells. The study also uses radiation, because laboratory and animal studies show that low doses of radiation to tumors that produce CEA make the tumor more sensitive to the effects of the vaccines.

Patients 18 years of age and older who have a solid tumor that has spread to the liver may be eligible for this study. Candidates must have had at least one course of chemotherapy for metastatic disease and their tumor must produce CEA. Candidates are screened with a medical history and physical examination; blood and urine tests, test of pathology slides from surgery to determine the presence of the CEA marker, imaging studies to assess the extent of tumor, and an electrocardiogram (and cardiologic evaluation, if clinically indicated).

Participants receive the priming vaccination on study day 1. After 3 weeks and then again every 2 weeks for 2 months (study days 21, 35, 49 and 63), they receive a boosting vaccine. All vaccines are injected under the skin. With every vaccination they also receive an injection of rF-GM-CSF to increase the number of immune cells at the vaccination site. The day after each of the first four boosting vaccinations, patients undergo 4 consecutive days of radiation to the tumor in the liver (study days 22-25, 36-39, 50-53 and 64-67). Patients may continue treatment with monthly booster vaccinations (without further radiation therapy) as long as their cancer does not get worse and they do not develop serious treatment side effects.

Patients are monitored for safety and treatment response with the following tests and procedures:

* Blood and urine tests and clinic visits every 2 to 4 weeks to monitor liver, kidney, and other organ function.
* Imaging studies to assess the tumor around study day 91 and every 2 months after that while on the study.
* Apheresis (a procedure for collecting immune cells called lymphocytes) - Apheresis is done before the first vaccination on study day 1 and again around study day 91. For this procedure, blood is collected through a needle in an arm vein. The blood circulates through a machine that separates it into its components by spinning, and the lymphocytes are extracted. The rest of the blood is returned to the patient through the same needle. The collected lymphocytes are studied to measure the immune response to treatment.
* Liver biopsy (optional) - This test is done once before starting radiation treatment and again around 3 to 7 days after completing the first dose of radiation. The biopsy provides information on the type of cancer, the level of CEA produced by the tumor, and the immune status of the tumor. For this procedure, the skin over the liver is numbed with an anesthetic, a needle is placed in the liver tumor, and a small sample of tumor is withdrawn through the needle.

After treatment is completed, patients are monitored for up to 15 years, including yearly medical histories and physical examinations for 5 years following their last vaccination. Information beyond 5 years is collected once a year by telephone

DETAILED DESCRIPTION:
Background:

* A phase I clinical trial with this same vaccine alone was associated with stable disease (at least 4 months) in 40% of patients and 1 pathologic complete response.
* Radiation therapy upregulates Fas on tumor cells allowing for easier killing by antigen specific activated T cells. Dominant negative fas transfected tumor cells demonstrated the anti-tumor effects were fas mediated.
* Radiation has been shown to up-regulate ICAM, tumor associated antigens and MHC class I on human tumor cell lines in vitro.
* TRICOM vaccines act synergistically with radiation in tumor treatment models.
* Radiation therapy at the doses we propose appears to have a favorable safety profile.
* Clinical trials using PSA vaccine shows that local radiation of tumor does not inhibit vaccine efficacy.

Objectives:

* 1: Safety of the combination of a CEA based vaccine and radiation
* 2: clinical response
* 2: Immunohistochemistry - (FAS, MHC, p53 and CEA on tumor before and after radiation therapy)
* 2: Immunological response (ELISPOT assay).

Eligibility:

* Solid Tumors expressing CEA positive cancer with radiographically visible metastatic liver lesions.
* Completed at least one chemotherapy regimen for metastatic disease.
* Life expectancy greater than or equal to 6 months
* Adequate organ function
* ECOG 0-1
* No autoimmunity
* No serum positivity for HIV, Hepatitis B or C viruses

Design:

* Single cohort pilot study of vaccine and radiation therapy to liver lesions in 10 evaluable patients. All vaccines and radiation are given at the NIH Clinical Center.
* Vaccine:

rV-CEA(6D)/TRICOM, (1.2 x 10(8)) PFU subcutaneously (s.c.) day 1

rF-CEA(6D)/TRICOM, (4 x 10(8)) PFU s.c., days 21, 35, 49, and 63

All vaccinations will be given with rF-GM-CSF, 1 x 10(7) pfu s.c.

-Radiation: 2 Gy/d for 4 days after each dose of rF-CEA(6D)/TRICOM on days 22-25, 36-39, 50-53, and 64-67 (total planned radiation dose per patient is 32 Gy).

ELIGIBILITY:
* INCLUSION CRITERIA

Solid Tumors expressing CEA positive cancer with radiographically visible metastatic liver lesions. Tumor that has been shown to express CEA by positive immunohistochemical techniques (staining of at least 20% of cells will be considered positive) or have had an elevated serum CEA greater than 5 ng/ml at any point during their disease course.

Completed at least one chemotherapy regimen for metastatic disease.

18 years of age or greater.

Life expectancy greater than or equal to 6 months.

Able to understand and give informed consent.

ECOG performance status of 0 - 1.

Serum creatinine within the institution limits of normal OR creatinine clearance on a 24 hour urine collection of greater than or equal to 60 mL/min, AST less than or equal to twice the institution upper limits of normal.

Total bilirubin less than the upper level of normal for that particular institution and if patient has Gilbert's syndrome, is bilirubin less than or equal to 3.0.

Vaccinia-naive or vaccinia immune.

Recovered completely from any reversible toxicity associated with recent therapy. Typically this is 3-4 weeks for patients who most recently received cytotoxic therapy except for the nitrosoureas and mitomycin C for which 6 weeks is needed for recovery.

At least 4 weeks after cytotoxic therapy with complete recovery of reversible toxicity.

Hematological eligibility parameters (within 16 days of starting therapy):

Granulocyte count greater than or equal to1,500/mm(3).

Platelet count greater than or equal to 100,000/mm(3).

Hgb greater than or equal to 8 Gm/dL.

Absolute lymphocyte count greater than or equal to 400/mm(3).

PT/PTT within the institution limits of normal.

Prior Immunotherapy will be allowed

Serum Beta-HCG less than 5.0 microIU/mL in females (with child bearing potential).

EXCLUSION CRITERIA

Patients should have no evidence of being immunocompromised as listed below.

* Human immunodeficiency virus positivity due to the potential for decreased tolerance and may be at risk for severe side effects
* Autoimmune diseases such as, Addison's disease, Hashimoto's thyroiditis, or systemic lupus erythematous, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome active Grave's disease. Altered immune function in prospective participants will be assessed through a thorough history and physical examination. Any clinical suspicion of autoimmune dysfunction will be worked up before enrollment on to the study. This requirement is due to the potential risks of exacerbating autoimmunity
* Hepatitis B or C positivity
* Prior radiation to greater than 50% of all nodal groups
* Prior whole liver radiation
* Concurrent use of systemic steroids, except for physiologic doses for systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Steroid eye drops are contraindicated for at least 2 weeks prior vaccinia vaccination and at least 4 weeks post vaccinia vaccination.
* Prior splenectomy

History of allergy or untoward reaction to prior vaccination with vaccinia virus or to any component of the vaccinia vaccine regimen.

Pregnant or breast-feeding women.

Recombinant vaccinia vaccination should not be administered if any of the following apply to either recipients, or for at least three weeks after vaccination (i.e., until the scab has separated from the skin and the underlying skin has healed), their close household contacts (close household contacts are those who share housing or have close physical contact): persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 5 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV infection.

Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.

Known brain metastasis, history of seizures, encephalitis, or multiple sclerosis.

Concurrent chemotherapy.

Serious hypersensitivity reaction to egg products.

Clinically significant cardiomyopathy requiring treatment.

Patients with cardiac disease that have fatigue, palpitation, dyspnea or angina with ordinary physical activity (New York Heart Association class 2 or greater) are not eligible.

Patients with pulmonary disease that have fatigue or dyspnea with ordinary physical activity are not eligible.

Patients who have objective evidence of congestive heart failure by physical exam or imaging are not eligible.

Chronic liver disease including end stage cirrhosis, or chronic active hepatitis as indicated by surface antigen or core antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-04-20; Primary Completion 2007-08-23 (Actual); Study Completion 2007-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahlers CM, Camphausen K, Citrin D, Arlen PM, Gulley JL. A pilot trial of a carcinoembryonic antigen/ TRICOM-based vaccine and radiation to liver metastases in patients with carcinoembryonic antigen-positive solid tumors. Clin Colorectal Cancer. 2006 May;6(1):72-5. doi: 10.3816/CCC.2006.n.025. No abstract available. PMID 16796796
- [Background] Ferrara TA, Hodge JW, Gulley JL. Combining radiation and immunotherapy for synergistic antitumor therapy. Curr Opin Mol Ther. 2009 Feb;11(1):37-42. PMID 19169958
- [Background] Hodge JW, Guha C, Neefjes J, Gulley JL. Synergizing radiation therapy and immunotherapy for curing incurable cancers. Opportunities and challenges. Oncology (Williston Park). 2008 Aug;22(9):1064-70; discussion 1075, 1080-1, 1084. PMID 18777956
- [Derived] Huang J, Jochems C, Talaie T, Anderson A, Jales A, Tsang KY, Madan RA, Gulley JL, Schlom J. Elevated serum soluble CD40 ligand in cancer patients may play an immunosuppressive role. Blood. 2012 Oct 11;120(15):3030-8. doi: 10.1182/blood-2012-05-427799. Epub 2012 Aug 28. PMID 22932804